CLINICAL TRIAL: NCT07215676
Title: An Open-Label Pilot Trial of a Multi-Component Nutritional Supplement in Hydrogen-Dominant Small Intestinal Bacterial Overgrowth
Brief Title: A Trial of a Multi-Component Nutritional Supplement in Hydrogen-Dominant Small Intestinal Bacterial Overgrowth
Acronym: AV1-SIBO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Natural Medicine (Other)
Responsible Party: Principal Investigator, Brice Thompson, Principal Investigator, National University of Natural Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: JG72425
Record Dates: First submitted 2025-09-16; First posted 2025-10-10 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Small Intestinal Bacterial Overgrowth Syndrome (SIBO); Small Intestinal Bacterial Overgrowth
Keywords: SIBO; small intestinal bacterial overgrowth; hydrogen SIBO; dysbiosis; probiotic; postbiotic
MeSH Terms: conditions — Dysbiosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AV1PD1A (Experimental): Multi-component dietary supplement taken 3 capsules daily for 8 weeks
  Interventions: Dietary Supplement: AV1PD1A

INTERVENTIONS:
Dietary Supplement: AV1PD1A — Saccharomyces cerevisiae fermentate, N-acetyl-glucosamine, Saccharomyces boulardii, heat-killed Lactobacillus rhamnosus, methylcobalamin, berberine, ginger extract

SUMMARY:
The goal of this trial is to evaluate the safety and tolerability of an 8-week, multi-component nutritional supplement (AV1PD1A) in adults with hydrogen-dominant small intestinal bacterial overgrowth (SIBO).

The main questions the study aims to answer are:

1. Is the product safe and well-tolerated over 8 weeks, as measured by bloodwork, vital signs, and adverse effects?
2. How many participants adhere to the intervention without a dose modification, hold, or discontinuation?

Exploratory questions include: do GI symptoms and quality of life ratings improve, and do hydrogen/methane levels on lactulose breath testing change from baseline to week 8?

There is no comparison group; this is a prospective, open-label, single-arm pilot trial (n=10).

Participants will:

* Be screened and confirmed to have hydrogen-dominant SIBO by lactulose breath test (with 24-hour prep diet and overnight fast).
* Take AV1PD1A, three capsules daily for 8 weeks.
* Attend three clinic visits at baseline, week 4, and week 8 for vital measurements, fasting blood draws, and adverse event checks.
* Complete questionnaires on symptoms and quality of life.
* Repeat the lactulose breath test at week 8 to assess changes in hydrogen and methane.

DETAILED DESCRIPTION:
Prospective, single-site, open-label, single-group pilot conducted at NUNM's Helfgott Research Institute (Portland, OR). The investigational product (AV1PD1A) is a multi-component dietary supplement containing Saccharomyces cerevisiae fermentate (EpiCor), N-acetyl-glucosamine, Saccharomyces boulardii, Lactobacillus rhamnosus (heat-killed), methylcobalamin, berberine, and gingerol (ginger extract). Dosing: 3 capsules daily for 8 weeks. Primary outcome is safety/tolerability (labs, vitals, AEs). Exploratory outcomes include validated PROMIS instruments, IBS Adequate Relief, and changes in lactulose breath-test hydrogen/methane. Enrollment is single-arm with anticipated n = 10 (pilot) to establish feasibility/tolerability signals that inform future powered trials.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 years.
* Meets North American Consensus criteria for hydrogen-dominant SIBO by lactulose breath test.
* Willing to: take study supplement (3 caps/day for 8 weeks); complete two lactulose breath tests with required prep/fast; undergo three fasting blood draws; complete questionnaires.
* Able to provide informed consent and communicate in English.
* Individuals of child-bearing potential agree to use effective contraception during the study.

Exclusion Criteria:

* Recent antibiotics/antifungals/supplements that confound breath test results (e.g., antibiotics within 14 days before breath test; current systemic or topical antifungals).
* Recent changes in diet/medications/supplement regimen within 30 days.
* Hospitalization within past 3 months.
* Allergy/intolerance to product components (e.g., Saccharomyces, Lactobacillus, shellfish [for N-acetyl-glucosamine], ginger, or berberine).
* Renal/hepatic abnormalities at screening (e.g., eGFR <60 mL/min/1.73 m2; AST/ALT/bilirubin outside of normal reference ranges).
* Hepatitis from any cause; excessive alcohol use (>7 drinks/week women; > 14 drinks/week men).
* Medications with concerning interactions after clinical investigator review

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-emergent adverse events any grade, per CTCAE v5.0 (Common Terminology Criteria for Adverse Events) | From baseline/enrollment to the end of treatment at 8 weeks
  The number of participants experiencing ≥1 treatment-emergent AE from first dose through end of treatment. Severity graded using CTCAE v5.0 (scale 1-5; 1 is least severe, 5 is most); relatedness assessed by the investigator. Report number of participants with any treatment-emergent AE and summarize by worst grade and relatedness.
Number of participants with laboratory abnormalities meeting pre-specified hold/stop criteria | Screening/baseline, Week 4, and Week 8
  Count of participants who meet any lab-based stopping rule (e.g., ALT/AST ≥3× ULN, total bilirubin ≥2× ULN, ALP ≥2× ULN with cholestatic pattern, eGFR <60 mL/min/1.73 m² on repeat or ≥50% decline from baseline, ANC <1,000/µL, Hgb <8 g/dL, platelets <50,000/µL). ULN/LLN per local lab report.
Number of participants requiring any dose modification/temporary hold/discontinuation | From first dose (Week 0) through end of treatment at Week 8.
  Count of participants who undergo a dose reduction, temporary hold, or permanent discontinuation of the study product per the prespecified dose-modification algorithm (triggered by AEs or labs).
Change in Patient Reported Outcomes Measurement Information System (PROMIS)-29+2 Profile v2.1 domain T-scores | From baseline/enrollment to the end of treatment at 8 weeks
  T-scores range from 22.5 minimum to 79.4 maximum. For symptom domains (e.g., Pain Interference, Anxiety, Depression, Fatigue, Sleep Disturbance), higher scores = worse symptoms; for function domains (Physical Function; Ability to Participate in Social Roles and Activities), higher scores = better function. Outcome is a mean change from baseline to Week 8 for the specified single domain.

SECONDARY OUTCOMES:
Change in PROMIS Gastrointestinal Gas & Bloating Short Form 6a T-score | From baseline/enrollment to the end of treatment at 8 weeks
  T-score range 20-80; higher = worse gas/bloating. Outcome is mean change from baseline to Week 8.
Change in PROMIS® Gastrointestinal Belly Pain Short Form 6a T-score | From baseline/enrollment to the end of treatment at 8 weeks
  T-score range 20-80; higher = worse belly pain. Outcome is mean change from baseline to Week 8.
IBS-Adequate Relief (IBS-AR) | From baseline/enrollment to week 4, to the end of treatment at 8 weeks.
  Proportion reporting adequate symptom relief at Week 4 and Week 8. The scale is a single dichotomous (yes/no) outcome from the question "Over the past week have you had adequate relief of your IBS symptoms?"
Change in 0-90-minute hydrogen rise (ppm) on lactulose breath test | From baseline/enrollment to the end of treatment at 8 weeks
  Mean change in 0-90 min hydrogen rise (ppm) from baseline to Week 8.
Change in peak methane (ppm) on lactulose breath test | From baseline/enrollment to the end of treatment at 8 weeks
  Mean change in peak methane (ppm) from baseline to Week 8. (Consensus: ≥10 ppm at any time indicates methane-positive.)
Number of participants with a negative lactulose breath test at Week 8 | Week 8
  Count of participants meeting negative criteria at Week 8 (e.g., hydrogen rise <20 ppm (0-90 min) and methane <10 ppm at all time points), per consensus thresholds.

CONTACTS AND LOCATIONS:
Locations (1):
- NUNM - Helfgott Research Institute, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No
Aggregate, de-identified results will be disseminated; IPD may be considered upon reasonable request and IRB/DUA approvals